CLINICAL TRIAL: NCT02839057
Title: Survival After Surgical Treatment of Axis Fractures in Elderly: A National Registry Based Cohort Study
Brief Title: Survival After Surgical Treatment of Axis Fractures in Elderly
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: AxisFractureSweden
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Spinal Fractures
Keywords: Axis fractures; Elderly; Mortality; Surgical treatment
MeSH Terms: conditions — Spinal Fractures | interventions — Conservative Treatment; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical treatment: Patients ≥70 years with C2 fracture coded in patient registry (ICD-10: S12.1) treated with surgical fracture stabilisation
  Interventions: Procedure: Surgical treatment
- Non-surgical treatment: Patients ≥70 years with C2 fracture coded in patient registry (ICD-10: S12.1) treated non-surgically
  Interventions: Procedure: Non-surgical treatment

INTERVENTIONS:
Procedure: Non-surgical treatment — Cervical collar immobilisation for 12 weeks.
  Other Names: Conservative treatment
  Groups: Non-surgical treatment
Procedure: Surgical treatment — Stabilisation of C2-fracture by posterior fusion C1-C2, posterior fusion C2-C3, anterior fusion C2-C3 (no postoperative collar) or anterior screw osteosynthesis C2 (postoperative collar for 6 weeks).
  Groups: Surgical treatment

SUMMARY:
Fractures of the second cervical vertebra (C2) are the most common spinal fracture among the elderly. Non-surgical treatment comprises of cervical collar treatment for 12 weeks, while surgical treatment for elderly could mean posterior fixation C1-C2 without collar treatment or anterior screw osteosynthesis C2 with 6 weeks of collar treatment. A meta-analysis of retrospective studies has recently found an improved survival with surgical treatment. This national registry study is designed to estimate the survival of non-surgical and surgical treatment in a population-based cohort.

DETAILED DESCRIPTION:
The Swedish National Patient Registry (NPR) is hosted by the Swedish Agency of Health and Welfare and contains all patient contacts within Sweden with a coverage of >90% for orthopaedic diagnoses. Registered are main diagnosis and co-morbidity using the ICD-9 code until 1996 and from 1997 onward ICD-10 codes. Treatment is coded since 1996 using the Swedish classification of surgical procedures. Furthermore, information on hospitalisation time is available from the registry.

In the Swedish Cause of Death Registry (CDR) all deaths in Sweden are registered with date of death and cause of death. While date of death coverage is complete, the cause of death has only 46% agreement with the final hospital diagnosis.

All patients with the main diagnosis of C2 fracture (ICD-10: S12.1) treated between January 1st 1996 to December 31st 2014 are extracted from the NPR and merged with the CDR for incident deaths. Prior to data transmission, the Swedish Agency of Health and Welfare anonymised the individual personal identification numbers using a key which remained with the Agency.

Invalid age data will be excluded either due to missing entries or mismatch with date of death. Multiple admissions (cases with same identification number but more than 12 months between admissions) and duplicate entries (cases with same identification number) will be removed from the dataset, after valuable co-morbidity data from the duplicate entries were stored in the original record. Duplicate entries originate from separate recordings from each hospital if the patient is referred to a specialised hospital. Furthermore, primarily non-surgically treated cases with a change of treatment modality are registered as surgical patients. The registered hospitalisation time for these patients is the combined non-surgical and surgical in-hospital treatment period.

From each record the Charlson Comorbidity Index (CCI) is calculated. Using Swedish surgical procedure codes for spinal fusion ("NAG") and spinal osteosynthesis ("NAJ") patients receiving surgical treatment were marked, and the cohort divided into two groups receiving non-surgical or surgical treatment.

The age distribution differences of patients with C2-fractures treated surgically and non-surgically was visualised with a density distribution plot. A logit logistic regression analysis identified covariates of surgical treatment assignment and was presented with 95% confidence intervals (C.I.) and statistical probability p. Goodness-of-fit of the model was presented with pseudo-r2 according to McFadden.

Using the Kaplan-Meier method for non-surgical and surgical treatment mean survival, as well as survival rate at 3 months, 1 year, and 2 years was determined, and visualised using a Kaplan-Meier plot with 99% C.I. With the Cox proportional hazards regression method multiple covariates contributing to survival are entered and hazard ratio (HR) presented with 95% C.I. and probability p. As relevant covariates for survival besides surgical treatment age, gender, spinal cord injury, and CCI were identified. Since the assumption was that the medical advancement improved patient survival in general during the last decades, even year of admission was included as covariate in the model. In order to identify a cut-off age where a treatment modality is not associated anymore with greater survival the adjusted HR of a certain age and above was plotted over age with 95% C.I.

ELIGIBILITY:
Inclusion Criteria:

* C2-fracture
* Age ≥70 years

Exclusion Criteria:

* no C2-fracture
* Age <70 years

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: National patient registry extract with patients suffering from C2 fracture
Sampling Method: Non-Probability Sample
Enrollment: 6231 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Survival | Censored observational time (20 years)
  Survival as registered in Swedish National Cause of Death Registry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robinson Y, Robinson AL, Olerud C. Systematic review on surgical and nonsurgical treatment of type II odontoid fractures in the elderly. Biomed Res Int. 2014;2014:231948. doi: 10.1155/2014/231948. Epub 2014 Feb 10. PMID 24683543